CLINICAL TRIAL: NCT02336100
Title: Diagnostic Value of Flexible Spectral Imaging Color Enhancement (FICE) Plus Probe-based Confocal Laser Endomicroscopy (pCLE) for Minimal Change Esophageal Reflux Disease (MERD) Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, Rapat Pittayanon, MD, Gastrointestinal Unit, King Chulalongkorn Memorial Hospital, King Chulalongkorn Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: RP010
Record Dates: First submitted 2015-01-06; First posted 2015-01-12 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Diagnostic technique and procedure
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Endoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GERD patient (Experimental): 36 GERD patients without obviously abnormality were examined by FICE and then followed by pCLE to evaluate minimal change esophagitis
  Interventions: Device: Endoscopy (FICE and pCLE)
- Control (Experimental): 18 control patients were were examined by FICE and then followed by pCLE to evaluate minimal change esophagitis
  Interventions: Device: Endoscopy (FICE and pCLE)

INTERVENTIONS:
Device: Endoscopy (FICE and pCLE) — FICE is Flexible Spectral Imaging Color Enhancement and pCLE is probe-based Confocal Lase Endomicroscopy

SUMMARY:
Gastroesophageal reflux disease (GERD) patients without obvious mucosal break by endoscopy were examined by FICE, followed by confocal. Validity scores for MERD diagnosis were analyzed.

DETAILED DESCRIPTION:
Thirty-six patients with suspected MERD (positive GerdQ but normal conventional endoscopy) and eighteen asymptomatic control were recruited. The new FICE (EPX-4450HD) was performed at non-magnified, x50, and x100 zoom levels. The criteria for positive FICE were; A) triangular indentation, B) punctuate erythema, C) villiform mucosa, or D) increased number of capillary vessel. At the same session, pCLE was applied to count the number of intrapapillary capillary loops (IPCLs) by using more than 5 IPCLs in 500x500 micron area as a criterion for MERD diagnosis. The validity scores of both modalities and interobserever agreement of pCLE interpretation was assessed.

ELIGIBILITY:
Inclusion Criteria:

1. age more than 18 year old
2. no PPI therapy in previous 2 weeks and
3. no esophageal tumor or stenosis or history of esophageal surgery.

Exclusion Criteria:

1. bleeding tendency including decompensated cirrhosis, chronic kidney disease
2. long term antiplatelets or anticoagulants,
3. pregnancy or
4. history of fluorescein allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
MERD diagnosis from FICE plus pCLE. | 8 months
Interobserver agreement in pCLE for MERD diagnosis | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Rapat Pittayanon, MD, Principal Investigator — king
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Patum Wan, Thailand